CLINICAL TRIAL: NCT03978000
Title: A Randomized, Double Blind, Parallel-group, Placebo Controlled Study to Evaluate the Efficacy and Safety of IBP-9414 in Premature Infants 500-1500g Birth Weight in the Prevention of Necrotizing Enterocolitis - The Connection Study
Brief Title: IBP-9414 for the Prevention of Necrotizing Enterocolitis - The Connection Study
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Infant Bacterial Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IBP-9414-020
Record Dates: First submitted 2019-06-05; First posted 2019-06-06 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Necrotizing Enterocolitis
MeSH Terms: conditions — Enterocolitis, Necrotizing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IBP-9414 (Active Comparator)
  Interventions: Drug: IBP-9414
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IBP-9414 — Oral suspension
  Arms: IBP-9414
Drug: Placebo — Sterile water
  Arms: Placebo

SUMMARY:
IBP-9414 will be evaluated in preterm infants with a birth weight of 500-1500g, compared to placebo with regards to efficacy and safety in the prevention of necrotizing enterocolitis.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age at birth of 23 weeks+0 days to 32 weeks+0 days
* Birth weight 500-1500g
* ≤ 48 hours of age
* Written informed consent from the subject´s legally authorized representative (LAR)

Exclusion Criteria:

* Participation in any other interventional clinical trial
* Infants in extremis to whom no further intensive care is offered by attending neonatologist
* Infants with, or at a high probability for, early onset sepsis
* Infants with recognized chromosomal anomalies
* Congenital or acquired gastrointestinal disease
* Earlier or planned administration of formulas, foods or supplements that contain added live bacteria
* Infants with known positive maternal HIV status

Max Age: 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2158 (Actual)
Dates: Start 2019-07-04 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Confirmed necrotizing enterocolitis (NEC) | From the first dose until the infant reaches 34 weeks + 6 days post-menstrual age
Time to sustained feeding tolerance | From the first dose until the infant reaches 34 weeks + 6 days post-menstrual age

SECONDARY OUTCOMES:
At least one clinical sign of NEC as reported by the investigator AND abdominal X-ray evidence of intestinal pneumatosis and/or portal venous gas confirmed by independent adjudication. | From the first dose until the infant reaches 34 weeks + 6 days post-menstrual age
Surgery (or autopsy) with confirmation of NEC | From the first dose until the infant reaches 34 weeks + 6 days post-menstrual age
Death all causes | From the first dose until the infant reaches 34 weeks + 6 days post-menstrual age
Number of days of hospitalization | From the first dose until the infant reaches 34 weeks + 6 days post-menstrual age
Weight gain in g/kg | Weeks 3 and 4 of age
Number of subjects growing at ≥100 g/kg/week | Weeks 3 and 4 of age
Days with clinical signs of feeding intolerance | From the first dose until the infant reaches 34 weeks + 6 days post-menstrual age

CONTACTS AND LOCATIONS:
Overall Officials: Josef Neu, MD, Principal Investigator — University of Florida College of Medicine, Gainsville, FL
Locations (89):
- United States (54):
  - Banner University Medical Center / University of Arizona, Tucson, Arizona
  - Arkansas Children'S Hospital, Little Rock, Arkansas
  - University of Arkansas For Medical Services, Little Rock, Arkansas
  - Loma Linda University Children Hospital, Loma Linda, California
  - Good Samaritan Hospital, Los Angeles, California
  - LAC & USC Medical Center, Los Angeles, California
  - University of Califorina, Los Angeles (UCLA), Los Angeles, California
  - Valley Childrens Hospital, Madera, California
  - Sharp Memorial Hospital, San Diego, California
  - St. Francis Medical Center, Colorado Springs, Colorado
  - Connecticut Children'S Medical Center - Uconn - School of Medicine, Hartford, Connecticut
  - University of Florida Health, Gainesville, Florida
  - Wolfson Children'S Hospital, Jacksonville, Florida
  - Uf Health Jacksonville, Jacksonville, Florida
  - University of Miami/Holtz Children'S Hospital, Miami, Florida
  - Sheridan Clinical Research / Plantation General Hospital, Plantation, Florida
  - University of South Florida, Tampa, Florida
  - St. Joseph'S Women'S Hospital, Tampa, Florida
  - Georgia Regents University, Augusta, Georgia
  - Children'S Hospital of the University of Illinois, Chicago, Illinois
  - North Shore University Health System, Evanston, Illinois
  - SIU School of Medicine - HSHS St. John's Children's Hospital, Springfield, Illinois
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Wesley Medical Center, Wichita, Kansas
  - Tufts Children's Hospital, Boston, Massachusetts
  - Harvard Medical School - Beth Israel Deaconess Medical Center (Bidmc), Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - C.S Mott Children'S Hospital, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Helen DeVos Children's Hospital Spectrum Health Research, Grand Rapids, Michigan
  - Children'S Minnesota, Minneapolis, Minnesota
  - Associates in Newborn Medicine - Saint Paul, Saint Paul, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Kings County Hospital Center, Brooklyn, New York
  - Cohen Children'S Medical Center of Ny, New Hyde Park, New York
  - Northwell Health Cohen Children'S Medical Center of Ny, New York, New York
  - Children'S Hospital At Montefiore, The Bronx, New York
  - Maria Fareri Children's Hospital - Westchester Medical Center, Valhalla, New York
  - Duke University, Durham, North Carolina
  - New Hanover Regional Medical Center, Wilmington, North Carolina
  - Wake Health Forest Baptist Health, Winston-Salem, North Carolina
  - Children'S Hospital At Ou Medicine, Oklahoma City, Oklahoma
  - Geisinger Health, Danville, Pennsylvania
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Jackson Madison County General Hospital, Jackson, Tennessee
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - St David'S Health Care - St. David'S Medical Center/North Austin Medical Center, Austin, Texas
  - University of Texas Medical Branch - Ocr, Galveston, Texas
  - Texas Health Presbyterian Hospital - Plano, Plano, Texas
  - Sheridan Healthcare of Texas, P.A./Medical City Plano, Plano, Texas
  - North Central Baptist Hospital, San Antonio, Texas
  - Children's Hospital of Richmind at VCU, Richmond, Virginia
  - West Virginia University Medical Center, Morgantown, West Virginia
- Bulgaria (5):
  - University Multiprofile Hospital for Active Treatment "Dr. Georgi Stranski" - Clinic of Neonatology, Pleven
  - University Multiprofile Hospital for Active Treatment, Plovdiv
  - Acibadem City Clinic Tokuda Hospital (Tokushukai Medical Corporation - Tokuda Hospital Sofia) (THS), Sofia
  - Specialized Hospital in Active Treatment of Pediatric Diseases, Sofia
  - University Hospital of Obstetrics and Gynecology Maichin Dom - Neonatology Clinic, Sofia
- France (3):
  - Chu Amiens-Picardie - Site Sud, Amiens
  - Centre Hospitalier Universitaire de Caen Normandie, Caen
  - Hopital Louis Mourier, Colombes
- Hungary (7):
  - University of Debrecen Clinical Center, Debrecen
  - Bács-Kiskun County Hospital, Kecskemét
  - Borsod- Abaúj-Zemplén County Central Hospital and University Teaching Hospital, Miskolc
  - Szszb County Hospital and Jósa András University Teaching Hospital, Nyíregyháza
  - University of Szeged, Albert Szent-Györgyi Health Centre, Szeged
  - Szent György University Teaching Hospital of County Fejér, Székesfehérvár
  - Veszprém County Csolnoky Ferenc Hospital, Veszprém
- Israel (3):
  - Carmel Medical Center, Haifa
  - Rambam Hospital, Haifa
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
- Poland (4):
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 Pomorskiego Uniwersytetu Medycznego im. prof. Tadeusza Sokołowskiego, Szczecin
  - Samodzielny Publiczny Szpital Kliniczny nr 2 Pomorski Uniwersytet Medyczny (PUM) w Szczecinie /Pomeranian Medical University, Szczecin
  - Uniwersyteckie Centrum Kliniczne, Warszawskiego Uniwersytetu Medycznego, Warsaw
  - Uniwersytecki Szpital Kliniczny, Wroclaw
- Romania (5):
  - Spitalul Clinic de Obstetrica si Ginecologie "Filantropia", Bucharest
  - Spitalul Clinic Judetean de Urgenta Cluj-Napoca, Cluj-Napoca
  - Spitalul Clinic de Obstetrica-Ginecologie "Cuza-Voda" Iasi, Iași
  - Spitalul Clinic de Urgenta pentru Copii "Louis Turcanu" Timisoara, Timișoara
  - Spitalul Clinic Municipal de Urgenta Timisoara, Timișoara
- Children's Clinic of the Clinical Center of Kragujevac, Kragujevac, Serbia
- Spain (5):
  - Hospital General de Alicante, Alicante
  - Hospital Clinico San Carlos - Idissc, Madrid
  - Hospital Universitario Hm Puerta Del Sur, Madrid
  - Hospital Juan XXIII, Tarragona
  - Hospital Universitario La Fe, Valencia
- United Kingdom (2):
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Nottingham University Hospitals, Neonatology: City Campus, Nottingham